CLINICAL TRIAL: NCT04818112
Title: A Randomized Controlled Trial to Improve Mother-Infant Synchrony Among Women With Childhood Adversity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Children's Wisconsin (Unknown)
Responsible Party: Principal Investigator, Aleeca Bell, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009050756
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Parent-Child Relations; Maternal Behavior; Infant Behavior
Keywords: Oxytocin; DNA methylation; Massage; Mothers; Infant; Adverse childhood experiences; Mother-infant interaction; Maternal behavior; Infant behavior; Receptor, oxytocin; Randomized controlled trial
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial uses group comparison of an intervention group and an education control group.
Who Masked: Outcomes Assessor
Masking Description: The video coders measuring mother-infant synchrony will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral ATVV intervention (Experimental): A multi-sensory behavioral intervention that includes auditory, tactile, visual and vestibular (ATVV) stimulation contingent upon infant cues.
  Interventions: Behavioral: ATVV
- Attention control (Active Comparator): An attention control group that receives education on safe infant care and the same amount of attention as the intervention group.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: ATVV — A 15-minute behavioral intervention that mothers administer once daily to their infant for 3 months providing Auditory, Tactile, Visual, and Vestibular (ATVV) stimulation. Multisensory stimuli are presented in gradual progression. Mother-infant engagement is attempted throughout ATVV so that mothers learn to identify, interpret and adapt to their infants cues. ATVV can be given without eye to eye gaze making it appropriate for newborns. ATVV is offered contingent on infant cues to promote self-regulation and withdrawn if any persistent disengagement cues. Mothers are taught how to adapt ATVV as their infant grows. Fidelity to the intervention is checked with weekly phone calls and monthly study visits. Mothers also receive a daily text from REDCap to document an intervention frequency log.
  Other Names: multisensory infant massage plus
  Arms: Behavioral ATVV intervention
Behavioral: Attention control — Mothers in the Attention Control group receive a similar amount of daily texts, weekly phone call and in-person study visit attention as mothers in the ATVV group, but with distinctly different content. Over the first 3 postnatal months, mothers learn safe infant-care that includes content on diapers, infant clothing, blankets, infant care including bathing, sleep positions, sleep habits, holding the baby, safety of infant equipment, breastfeeding, formula, and age appropriate toys.
  Arms: Attention control

SUMMARY:
Childhood adversity affects almost two-thirds of the US population, is a major risk factor for the leading causes of disease and increases US economic health burdens. Childhood adversity also alters biologic systems, such as the oxytocin hormone, that can affect attachment behavior. This innovative study has the potential to advance science and improve mother-infant interaction by testing an early life, home-based, multisensory behavioral intervention (called ATVV), targeting the oxytocin system, to promote synchronous early mother-infant interaction, especially critical for mothers who have experienced childhood adversity.

This two-group randomized clinical trial will test the ATVV's effect on oxytocin system function and quality of mother-infant interaction. The investigators will enroll 250 first-time healthy mothers carrying a single baby who have a history of childhood adversity, and obtain baseline data in their third trimester of pregnancy. Soon after birth (before hospital discharge), mothers (and babies) who continue to be eligible are randomized into the intervention group and taught to give ATVV daily for 3 months, or randomized into the Attention Control education group and taught safe infant care. After birth, the investigators check-in frequently with mothers through weekly phone calls. There are 3 study visits at 1, 2 and 3 months after birth that include survey questions and collection of maternal blood and infant saliva. Mothers and babies are also video-recorded at 3 months after birth for 4 minutes to assess mother-infant interaction. The investigators follow-up with a phone call at 6 months after birth.

While both groups will benefit from the content and attention the investigators give mothers, the investigators hypothesize that, compared to the education group, mothers and infants in the intervention group will have improved oxytocin system function and more synchronous mother-infant interaction.

DETAILED DESCRIPTION:
Childhood adversity (e.g., abuse, neglect, or household dysfunction), is a common experience significantly contributing to the leading causes of death and increased US economic health burdens. Childhood adversity causes long-term alterations on the nervous, endocrine, and immune systems well into adulthood, including dampening of the neuropeptide oxytocin (OXT). A healthy OXT system facilitates responsive social engagement and promotes maternal-infant (M-I) synchrony (reciprocal gaze, affect speech, and touch). Optimal M-I synchrony fuels early brain development and prevents low empathy, disruptive behavior, poor social adaptation, cognitive deficits, and psychopathology in children. The investigators posit that mothers with childhood adversity will have more difficulty with M-I synchrony, due in part to a dampened OXT system, and will benefit from interventions that improve responsive, nurturing, engagement by epigenetic regulation of the OXT system. Most interventions are costly, complex, and time-consuming. The investigators aim to fill this gap by testing whether a simple early behavioral intervention (ATVV) will improve OXT system function and M-I synchrony in mothers with childhood adversity.

The ATVV (Auditory, Tactile, Visual, Vestibular) is a 15-minute behavioral intervention that is a multisensory infant massage contingent on infant cues. The investigators extend the known success of ATVV with preterm infants to full-term infants. The investigators will compare M-I synchrony at 3 postnatal months in 250 first-time mothers (and their full-term infants) randomized to apply ATVV daily from birth to 3 months (n =125) or receive infant care education in an attention control group (n = 125). The investigators apply a rigorous measure of M-I synchrony that micro-codes video-recorded M-I behavior quantifying shared gaze, affect, speech, and touch. Coding requires only 3-minutes of interaction and is valid when infants can reliably interact starting by 3 months of age. The investigators will also assess ATVV's effect on maternal and infant peripheral OXT level, a known biomarker of M-I synchrony. OXT levels relate to quality of M-I synchrony, yet the investigators extend this knowledge to identify an epigenetic role of the oxytocin receptor gene (OXTR). The investigators will analyze maternal plasma for OXTR methylation, OXTR gene expression, OXTR protein, and oxytocin peptide in pregnancy, and at 1, 2, and 3 postnatal months (along with infant saliva OXT).

The investigators propose a single-site, randomized, two-group, attention-controlled clinical trial (N=250 M-I dyads) to test the efficacy of the ATVV multisensory behavioral intervention to improve OXT system function and M-I synchrony. Adult, nulliparous, English or Spanish speaking women carrying a single fetus, and scoring 2 or higher on the Adverse Childhood Experiences scale will be enrolled. The investigators will obtain baseline OXT, demographics and survey data in the third trimester. Soon after birth (pre-hospital discharge), M-I dyads who continue to be eligible (e.g., full-term gestation) are randomized into the intervention group (n = 125) and taught to administer ATVV daily for 3 months or randomized into the Attention Control group (n = 125) and taught normal safe infant care. There are postnatal study visits at 1, 2 and 3 months. The investigators follow-up with a phone call at 6 postnatal months (3-months after the intervention period ends) to assess self-report parenting behavior (a proxy for quality of M-I interaction) that the investigators also measure at postnatal months 1, 2, and 3.

Aim 1: Evaluate the efficacy of daily ATVV over 3 postnatal months among mothers with childhood adversity. The investigators hypothesize that compared to the Attention Control group (n=125), M-I dyads in the ATVV group (n=125) will exhibit:

H1: Higher oxytocin function (i.e., decreased OXTR methylation at candidate sites, and increased OXTR messenger ribonucleic acid (mRNA), OXTR protein, and OXT in maternal plasma, and increased OXT in infant saliva) at 1, 2, and 3 postnatal months.

H2: More synchronous eye-to-eye gaze [primary], positive affect [primary], speech, and touch at 3 postnatal months.

Aim 2: Identify molecular mechanisms in the OXT system underlying M-I synchrony (N=250).

H1: Lower M-I synchrony will be associated with dampening of the OXT system, evidenced by increased OXTR methylation at candidate sites, and decreased OXTR mRNA, OXTR protein, and OXT in maternal plasma, and decreased OXT in infant saliva at 3-postnatal months.

Regression based methods (including covariates) will assess ATVV effects on M-I synchrony and OXT measures, and identify relations among M-I synchrony and oxytocin measures. Clustering methods will be used to discover molecular profiles. An early behavioral intervention that successfully promotes M-I synchrony in vulnerable women through epigenetic regulation of the OXT system can then be tested in a multi-site clinical implementation trial with other high-risk groups.

Protocol: The Recruiter will introduce the study to potentially eligible pregnant women. Eligible women who are interested in joining will be consented and scheduled for a 3rd trimester baseline study visit at the university. The investigators will draw blood for OXT measures, and collect data in REDCap on demographics, maternal characteristics, and self-report surveys. Research team members will keep track of when participants have given birth and meet them in a study site hospital before discharged. The investigators will collect data on mother and infant health, birth events, and other covariates. At the hospital visit, women are randomly assigned to either the ATVV group and taught how to administer the intervention on a daily basis, or are randomly assigned to the Attention Control group and taught safe infant newborn care.

All participants will receive daily texts to measure daily stress, and intervention participants also document frequency of the intervention. Using Participatory Guidance to address women's needs, the investigators will call women each week after birth for a check-in. In the intervention group, any challenges with the intervention will be discussed and problem-solved. In the Attention Control group, age-appropriate safe infant care will be discussed.

After the hospital visit, monthly study visits at 1, 2, and 3 months include collecting maternal blood and infant saliva, and self-report surveys in REDCap. Women will either complete REDCap surveys online before each visit, or complete them at the study visit. To check intervention fidelity, mothers in the ATVV group demonstrate how they perform the intervention with their infant. The team member instructs mothers how to adapt the ATVV to their maturing infant and discuss any challenges with the intervention. Mothers in the Attention Control group are taught age-appropriate safe infant care.

At the 3rd month study visit, the investigators collect behavioral outcome data on M-I synchrony. All M-I dyads will be video recorded freely interacting with each other for 4 minutes (coding occurs on the last 3 minutes). Video recording occurs when the infant is alert and ready to interact, > 30 minutes after the end of a breastfeeding or formula feeding, and data collection order may be adjusted if the baby is sleepy or fussy. Interactions are micro-coded frame by frame on a computerized system (Noldus, Wageningen, The Netherlands), consistent with previous research on parent-infant synchrony. Coders, blinded to group assignment, are trained to 90% inter-rater reliability. Our last interaction with participants is a phone call at 6-postnatal months to explore duration of the intervention's effect using the Parenting Stress Index.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant
2. Healthy (gestational diabetes is acceptable)
3. Greater than or equal to 18 years old
4. Nulliparous (previous miscarriage(s) and/or abortion(s) acceptable)
5. Speak and read English or Spanish
6. Score greater than or equal to 2 on the Adverse Childhood Experience (ACE) survey
7. Expect to deliver a healthy infant
8. Expect to deliver a full-term infant (greater than or equal to 37 weeks and 0/7 days)
9. Expect to deliver a singleton infant

Exclusion Criteria:

1. Multiparous
2. Have no access to a cell phone during the first 3 postnatal months
3. Carrying multiple fetuses
4. Taking anti-depressant(s) during pregnancy
5. Taking illicit drugs
6. Do not speak and read English or Spanish;
7. Under 18 years of age
8. Score less than 2 on the Adverse Childhood Experience (ACE) survey
9. Deliver an infant diagnosed with conditions that could affect normal development or the oxytocin system

   1. Pre-term gestation (less than 37 weeks and 0/7 days)
   2. Intrauterine growth retardation (IGR)
   3. Small for gestational age (SGA)
   4. Chromosomal anomaly including

      * Down syndrome (trisomy 21)
      * Trisomy 13
      * trisomy 18
      * Klinefelter syndrome
      * Turner syndrome
      * Triple X syndrome
   5. Congenital anomaly including

      * Heart defect
      * Musculoskeletal defect
      * Neural tube defect
      * Cystic Fibrosis
      * Haemophilia
      * Microcephaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleeca Bell, PhD, Principal Investigator — University of Arizona, College of Nursing
Locations (2):
- United States (2):
  - Tucson Medical Center, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (pregnant women) were consented prior to birth. The 262 consented pregnant women are the protocol enrollment number. Between consent and randomization, participants attended a baseline study visit and gave birth. During this period, 49 pregnant women or mother-infant dyads were excluded due to lost to follow-up, no longer meeting inclusion criteria, or withdrawal. Randomization reflects mother-infant dyads at birth: 107 dyads in the intervention, 106 dyads in the control.
Period: Overall Study
Arm/Group | Behavioral ATVV Intervention | Attention Control
Started | 214 (107 mothers and 107 infants) | 212 (106 mothers and 106 infants)
Completed | 122 (61 mothers and 61 infants) | 190 (95 mothers and 95 infants)
Not Completed | 92 | 22
Not completed — Withdrawal by Subject | 54 | 12
Not completed — Lost to Follow-up | 38 | 10

BASELINE CHARACTERISTICS:
Population: Participants included both mothers and infants. Two dyads withdrew after randomization prior to receiving the intervention, explaining the discrepancy between randomized and analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral ATVV Intervention | Attention Control | Total
Number analyzed (Participants) | 210 | 212 | 422
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants included both mothers and infants.
  Participants
    Mothers: number analyzed (Participants) | 105 | 106 | 211
    Mothers: <=18 years | 0 | 0 | 0
    Mothers: Between 18 and 65 years | 105 | 106 | 211
    Mothers: >=65 years | 0 | 0 | 0
    Infants (perinates): number analyzed (Participants) | 105 | 106 | 211
    Infants (perinates): <=18 years | 105 | 106 | 211
    Infants (perinates): Between 18 and 65 years | 0 | 0 | 0
    Infants (perinates): >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants included both mothers and infants.
  Participants
    Mothers: number analyzed (Participants) | 105 | 106 | 211
    Mothers: Female | 105 | 106 | 211
    Mothers: Male | 0 | 0 | 0
    Infants (perinates): number analyzed (Participants) | 105 | 106 | 211
    Infants (perinates): Female | 53 | 47 | 100
    Infants (perinates): Male | 52 | 59 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants included both mothers and infants.
  Participants
    Mothers: number analyzed (Participants) | 105 | 106 | 211
    Mothers: Hispanic or Latino | 50 | 53 | 103
    Mothers: Not Hispanic or Latino | 55 | 53 | 108
    Mothers: Unknown or Not Reported | 0 | 0 | 0
    Infants: number analyzed (Participants) | 105 | 106 | 211
    Infants: Hispanic or Latino | 50 | 53 | 103
    Infants: Not Hispanic or Latino | 55 | 53 | 108
    Infants: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants included both mothers and infants.
  Participants
    Mothers: number analyzed (Participants) | 105 | 106 | 211
    Mothers: American Indian or Alaska Native | 1 | 3 | 4
    Mothers: Asian | 4 | 5 | 9
    Mothers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Mothers: Black or African American | 4 | 3 | 7
    Mothers: White | 67 | 74 | 141
    Mothers: More than one race | 4 | 6 | 10
    Mothers: Unknown or Not Reported | 25 | 15 | 40
    Infants: number analyzed (Participants) | 105 | 106 | 211
    Infants: American Indian or Alaska Native | 1 | 3 | 4
    Infants: Asian | 4 | 5 | 9
    Infants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Infants: Black or African American | 4 | 3 | 7
    Infants: White | 67 | 74 | 141
    Infants: More than one race | 4 | 6 | 10
    Infants: Unknown or Not Reported | 25 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mother-Infant Synchrony, Gaze and Affect
Description: Video-recordings of mothers freely interacting with their infant were micro-coded second by second for the number of seconds of mother-infant synchrony over 180 seconds. Behaviors are categorized into mutually exclusive codes. The most robust behavior categories for mothers and infants (individually and in synchrony) are gaze and affect. Maternal gaze consisted of mother's gaze to infant's face, to infant's body, to object or environment, and gaze aversion. Infant gaze consisted of gaze to mother, gaze to object or environment, and gaze aversion. Maternal affect consisted of positive, neutral, and negative affective expression. Infant affect consisted of high positive (laugh, giggle, smile), positive (smile, bright face), negative (sad face, occasional whimper), high negative (cry, strong whining), or neutral.
Time Frame: 84 +/- 7days from birth (approximately 3 months after birth)
Population: This is the number of subjects at 3 months postpartum with video recordings to measure mother-infant synchrony. 64 dyads in the behavioral ATVV intervention were analyzed, and 98 dyads in the Attention Control were analyzed.
Measure: Mean (95% Confidence Interval); unit: seconds of synchrony
Arm/Group | Behavioral ATVV Intervention | Attention Control
Number analyzed (Participants) | 128 | 196
seconds of synchrony
  Gaze | 113.89 [103.58 to 124.20] | 106.72 [98.39 to 115.05]
  Affect | 28.2 [23.03 to 33.38] | 16.1 [11.92 to 20.29]

2. Secondary Outcome: Mother-Infant Synchrony, Vocalization and Touch
Description: Video-recordings of mothers freely interacting with their infant were micro-coded second by second for the number of seconds of mother-infant synchrony over 180 seconds. Behaviors are categorized into mutually exclusive codes. The second most robust behavior categories for mothers and infants (individually and in synchrony) are vocalization and touch. Maternal vocalization consisted of motherese positive speech (infant-directed speech typically high-pitched with a sing-song rhythm), adult speech to the infant in a normal range and regular rhythm, adult speech to other adult, and no speech. Infant vocalization consisted of positive (babbling, cooing, or giggles) and negative (fussing or crying).
Time Frame: 84 +/- 7days from birth (approximately 3 months after birth)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds of synchrony
Arm/Group | Behavioral ATVV Intervention | Attention Control
Number analyzed (Participants) | 128 | 196
seconds of synchrony
  Vocalization | 9.86 [7.28 to 12.44] | 9.76 [7.65 to 11.87]
  Touch | 16.05 [12.62 to 19.47] | 11.49 [8.72 to 14.26]

3. Secondary Outcome: Oxytocin Receptor Gene DNA Methylation Reflecting Epigenetic Marks
Description: Using maternal plasma, % OXTR DNA methylation will be measured at candidate cytosine-phosphate-guanosine (CpG) sites -1001, -959, -934, -924, -901, and -860 that were selected based on their implication in previous studies relating to psychosocial behaviors. There is also cost-effectiveness in using the selected assay to co-target additional CpG regions implicated in the literature relating to psychosocial behaviors. Methylation is measured using bisulfite conversion (EZ DNA Lightning Kit), followed by high-throughput next-generation sequencing of polymerase chain reaction (PCR) amplicons (Illumina MiSeq) at the University of Arizona Genetics Core.
Time Frame: Baseline at 31weeks +/- 2 weeks gestation and every 28 days +/- 7 days from birth to 3 months
Reporting Status: Not Posted, anticipated posting 2025-10

4. Secondary Outcome: Oxytocin Receptor Gene Expression
Description: Using maternal plasma, OXTR mRNA level will be measured using quantitative Real-Time PCR (qRT-PCR) that demonstrates total OXTR gene expression. This reflects the DNA transcribed (copied) into RNA before translation produces protein. Analysis is performed by the College of Nursing Biological Core Laboratory.
Time Frame: Baseline at 31weeks +/- 2 weeks gestation and every 28 days +/- 7 days from birth to 3 months
Reporting Status: Not Posted, anticipated posting 2025-10

5. Secondary Outcome: Oxytocin Receptor Protein
Description: Using maternal plasma, total protein expression of OXTR will be measured to reflect the amount of OXT receptors available to bind with OXT peptides. Analysis is performed by the College of Nursing Biological Core Laboratory using Anti-OXTR antibody and Western Blot (considered to be the gold standard).
Time Frame: Baseline at 31weeks +/- 2 weeks gestation and every 28 days +/- 7 days from birth to 3 months
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: Oxytocin Peptide, Maternal Plasma
Description: Using maternal plasma, the ELISA assay will be used to report OXT peptide level. Samples are analyzed at the University of Arizona Laboratory for the Evolutionary Endocrinology of Primates (LEEP) in duplicate by enzyme immunoassay (EIA) using the Oxytocin ELISA kit (Enzo; ADI-901-153A-0001).
Time Frame: Baseline at 31weeks +/- 2 weeks gestation and every 28 days +/- 7 days from birth to 3 months
Reporting Status: Not Posted, anticipated posting 2026-06

7. Secondary Outcome: Oxytocin Peptide, Infant Saliva
Description: Using infant saliva, the ELISA assay will be used to report OXT peptide level. Samples are analyzed at the University of Arizona Laboratory for the Evolutionary Endocrinology of Primates (LEEP) in duplicate by enzyme immunoassay (EIA) using the Oxytocin ELISA kit (Enzo; ADI-901-153A-0001).
Time Frame: Every 28 days +/- 7 days from birth to 3 months
Reporting Status: Not Posted, anticipated posting 2025-10

ADVERSE EVENTS:
Time Frame: From consent in pregnancy to 3 months after birth
Groups:
- Behavioral ATVV Intervention - Mothers; Behavioral ATVV Intervention - Infants: A multi-sensory behavioral intervention that includes auditory, tactile, visual and vestibular (ATVV) stimulation contingent upon infant cues.
  ATVV: A 15-minute behavioral intervention that mothers administer once daily to their infant for 3 months providing Auditory, Tactile, Visual, and Vestibular (ATVV) stimulation. Multisensory stimuli are presented in gradual progression. Mother-infant engagement is attempted throughout ATVV so that mothers learn to identify, interpret and adapt to their infants cues. ATVV can be given without eye to eye gaze making it appropriate for newborns. ATVV is offered contingent on infant cues to promote self-regulation and withdrawn if any persistent disengagement cues. Mothers are taught how to adapt ATVV as their infant grows. Fidelity to the intervention is checked with weekly phone calls and monthly study visits. Mothers also receive a daily text from REDCap to document an intervention frequency log.
- Attention Control - Mothers; Attention Control - Infants: An attention control group that receives education on safe infant care and the same amount of attention as the intervention group.
  Attention control: Mothers in the Attention Control group receive a similar amount of daily texts, weekly phone call and in-person study visit attention as mothers in the ATVV group, but with distinctly different content. Over the first 3 postnatal months, mothers learn safe infant-care that includes content on diapers, infant clothing, blankets, infant care including bathing, sleep positions, sleep habits, holding the baby, safety of infant equipment, breastfeeding, formula, and age appropriate toys.
Arm/Group | Behavioral ATVV Intervention - Mothers | Attention Control - Mothers | Behavioral ATVV Intervention - Infants | Attention Control - Infants
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/106 | 0/105 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/106 | 0/105 | 0/106
Other Adverse Events (participants affected / at risk) | 0/105 | 0/106 | 0/105 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT04818112/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT04818112/ICF_001.pdf